CLINICAL TRIAL: NCT03960827
Title: Molecular Transducers of Physical Activity Consortium
Acronym: MoTrPAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Stanford University (Other); Broad Institute of MIT and Harvard (Other); Duke University (Other); Emory University (Other); Icahn School of Medicine at Mount Sinai (Other); Pacific Northwest National Laboratory (U.S. Federal Agency); University of Michigan (Other); Wake Forest University (Other); University of Vermont (Other); National Institutes of Health (NIH) (NIH); National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH); Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB00097219; 1U24AR071113-01 (NIH); 5U24OD026629-03 (NIH); 1U24DK112349-01 (NIH); 1U24DK112342-01 (NIH); 1U24DK112340-01 (NIH); 1U24DK112341-01 (NIH); 1U24DK112326-01 (NIH); 1U24DK112331-01 (NIH); 1U24DK112348-01 (NIH); 1U01AR071133-01 (NIH); 1U01AR071130-01 (NIH); 1U01AR071124-01 (NIH); 1U01AR071128-01 (NIH); 1U01AR071150-01 (NIH); 1U01AR071160-01 (NIH); 1U01AR071158-01 (NIH)
Record Dates: First submitted 2018-03-26; First posted 2019-05-23 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2025-05

CONDITIONS: Physical Activity
Keywords: endurance exercise; resistance exercise; physical activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: The randomized trial is conducted in accordance with an intent-to-treat (ITT) design.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Sedentary control (No Intervention): The control group does not engage in any acute exercise testing protocol, but biospecimens are collected prior to and following a period of rest.
- Sedentary EE (Active Comparator): Participants randomized to EE first engage in a single acute exercise test of Endurance Exerciser (on a cycle ergometer) consistent with their random assignment.
  Interventions: Other: EE Training
- Sedentary RE (Active Comparator): Participants randomized to RE first engage in a single acute exercise test of Resistance Exerciser, consistent with their random assignment.
  Interventions: Other: RE Training
- Highly Active EE (No Intervention): A comparison group of highly active EE participants are recruited and engage only in the initial round of acute exercise testing. Highly Active Endurance Exerciser (HAEE) participants are tested on a cycle ergometer.
- Highly Active RE (No Intervention): A comparison group of highly active RE participants are recruited and engage only in the initial round of acute exercise testing. Highly Active Resistance Exerciser (HARE) participants are tested via a bout of resistance exercise.

INTERVENTIONS:
Other: EE Training — Participants randomized to EE engage in four center-based EE sessions each week for 12 weeks; each session lasting roughly 1-hour with a 40-45 minute stimulus phase and the remaining time being used to warm up and cool down. Each week, two of the sessions occur on a cycle ergometer and two involve treadmill exercise (4 total sessions per week). During all sessions, the participant's heart rate is monitored to ensure they maintain exercise intensity at 70% of heart rate reserve (± 5%). Periodically during training sessions perceptual data from participants are recorded, which is used to track the subjective experience of participants and in interpreting adherence data.
  Arms: Sedentary EE
Other: RE Training — Participants randomized to RE engage in four center-based RE sessions each week for 12 weeks; each session lasting roughly 1-hour with a 40-45 minute stimulus phase and the remaining time being used to warm up and cool down. The prescription is a 2-day split, meaning approximately half of the major muscle groups are exercised each session and each muscle group is exercised twice per week. Two sessions per week include seven exercises that focus on the hips/thighs, back and biceps, and the other two sessions per week include seven exercises that focus on the chest, shoulders, triceps, calves and abdominal muscles. The first set per muscle group is a warm-up performed at 50-70% of prescribed loads that are based on 10-repetition maximum (10RM). Three sets per exercise are then performed at 10RM intensity. Load increases when a participant can perform 12 repetitions for 2 of 3 sets of an exercise. During all sessions, heart rate is monitored and perceived exertion is recorded.
  Arms: Sedentary RE

SUMMARY:
The goal of the Molecular Transducers of Physical Activity Consortium (MoTrPAC) is to assess molecular changes that occur in response to physical activity (PA). To achieve this aim, a mechanistic randomized controlled trial (RCT) is conducted, in which adult study participants are randomized to endurance exercise (EE) training, resistance exercise (RE) training, or no exercise Control for a period of approximately 12 weeks. The overarching hypothesis is that there are discoverable molecular transducers that communicate and coordinate the effects of exercise on cells, tissues, and organs, which may initiate processes ultimately leading to the health benefits of exercise. Because this is a mechanistic trial, the main goal is not a single health-related outcome. Rather, the goal is to generate a resource leading to the generation of a map of the molecular responses to exercise that will be used by the Consortium and by the scientific community at large to generate hypotheses for future investigations of the health benefits of PA.

DETAILED DESCRIPTION:
Study assessments are completed before and after the intervention period (exercise or control), and at specific interim time points during the intervention. Assessments include measurements of cardiorespiratory fitness, muscular strength, and body composition (including total body bone mineral content) determined by dual-energy x-ray absorptiometry (DXA). There is also collection of blood, muscle, and adipose tissue biospecimens, monitoring of free-living PA level using wearable devices, and completion of participant reported outcomes and health status by interview and/or questionnaire. An additional group of highly active (HA) individuals currently active in either EE (HAEE) or RE (HARE) are recruited for a single acute exercise testing session of either endurance or resistance exercise and other study assessments. MoTrPAC participants are recruited, trained, and assessed via six adult Clinical Centers (CC), involving 10 clinical sites. As part of the MoTrPAC functions, participant data and biological samples are transferred from the clinical sites to the Consortium Coordinating Center (CCC) Data Management, Analysis and Quality Control Center (DMAQC)and to the Biological Sample Repository, and later analyzed by the Consortium Chemical Analysis Sites (CAS) and the Bioinformatics Center (BIC).

Biological samples collected in this project undergo molecular phenotyping, including metabolomic, lipidomic, proteomic, epigenomic, transcriptomic, and genomic analyses. These assays are done at the MoTrPAC CAS.

Overall coordination of the study and analyses occurs at 4 institutions which make up the CCC and the BIC.

ELIGIBILITY:
ADULT PARTICIPANT INCLUSION CRITERIA - SEDENTARY PARTICIPANTS

* Willingness to provide informed consent to participate in the MoTrPAC Study
* Must be able to read and speak English well enough to provide informed consent and understand instructions
* Aged ≥18 y
* Body Mass Index (BMI) ≥19 to ≤35 kg/m2
* Sedentary defined as self-reporting no more than 1 day per week, lasting no more than 60 minutes, of regular (structured) EE [e.g., brisk walking, jogging, running, cycling, elliptical, or swimming activity that results in feelings of increased heart rate, rapid breathing, and/or sweating] or RE (resulting in muscular fatigue) in the past year

  * Persons bicycling as a mode of transportation to and from work >1 day/week etc. are not considered sedentary
  * Leisure walkers are included unless they meet the heart rate, breathing, and sweating criteria noted above
  * Willingness to include de-identified individual-level data at low risk of re-identification (e.g.,non-genomic data) in the MoTrPAC open-access database
  * Only one member of a household can participate

ADULT PARTICIPANT INCLUSION CRITERIA - HIGHLY ACTIVE PARTICIPANTS

* Willingness to provide informed consent to participate in the MoTrPAC Study
* Must be able to read and speak English well enough to provide informed consent and understand instructions
* Aged ≥18 y
* BMI ≥19 to ≤35 kg/m2
* Comparator Participants

  * HAEE: defined as ≥240 minutes/week of ET for ≥1 year; this can include running, walking (brisk, power), cycling, elliptical, etc. which (at a minimum) results in increased heart rate, rapid breathing and sweating
  * Must include cycling at least 2 days/week
  * RT in the past year must be limited to ≤2 days/week of upper body RE and ≤2 muscle groups of upper body RE and ≤1 day/week of lower body RE
  * HARE: defined as RT of ≥3 upper and ≥3 lower body muscle groups ≥2 times/week for ≥1 year; using a prescription sufficient to increase strength and muscle mass
  * ET in the past year must be limited to ≤90 minutes/week of vigorous EE, with no limit on cycling days per week
  * Elite or Competitive Athletes: can be included, if they meet HAEE or HARE inclusion criteria
  * Potential participants are informed that use of performance enhancing drugs in the last 6 months is exclusionary
  * Willingness to include de-identified individual-level data at low risk of re-identification (e.g., non-genomic data) in the MoTrPAC open-access database
  * In addition to meeting HAEE or HARE inclusion criteria, all HA participants must meet all other exclusion criteria defined in this protocol

EXCLUSION CRITERIA

ADULT PARTICIPANT EXCLUSION CRITERIA Exclusion criteria are confirmed by self-report (i.e., medical and medication histories reviewed by a clinician), screening tests performed by the MoTrPAC study team at each clinical site, and/or clinician judgement as specified for each criterion.

* Diabetes (self-report and screening tests)

  * Treatment with any hypoglycemic agents (self-report) or A1c >6.4% (screening test; may reassess once if 6.5-6.7%)
  * Fasting glucose >125 mg/dL (screening test; may reassess once)
  * Use of hypoglycemic drugs for non-diabetic reasons (self-report)
* Abnormal bleeding or coagulopathy (self-report)

  * History of a bleeding disorder or clotting abnormality
* Thyroid disease (screening test)

  * Thyroid Stimulating Hormone (TSH) value >5.9 IU/mL
  * Individuals with hypothyroidism may be referred to their primary care provider (PCP) for evaluation and retested; any medication change must be stable for ≥3 months prior to retesting
  * Individuals with hyperthyroidism are excluded, including those with normal TSH on pharmacologic treatment
* Pulmonary (self-report)

  * Clinical diagnosis of Chronic Obstructive Pulmonary Disease (COPD)
* Metabolic bone disease (self-report)

  * History of non-traumatic fracture from a standing height or less
  * Current pharmacologic treatment for low bone mass or osteoporosis, other than calcium, vitamin D, or estrogen
* Estrogens, progestins (self-report)

  * Supplemental, replacement or therapeutic use of estrogens or progestins within the last 6 months, other than birth control or to control menopausal symptoms
* Pregnancy (screening test) and pregnancy-related conditions (self-report)

  * Pregnant - pregnancy test performed on day of DXA scan in women of child-bearing potential
  * Post-partum during the last 12 months
  * Lactating during the last 12 months
  * Planning to become pregnant during the participation period
* Elevated blood pressure readings (screening test)

  * Resting Systolic Blood Pressure (SBP) ≥150 mmHg or Resting Diastolic Blood Pressure (DBP) ≥95 mmHg
  * Reassessment of BP during screening will be allowed to ensure rested values are repeatable
* Cardiovascular (self-report, screening test, and clinician judgement)

  * Congestive heart failure, coronary artery disease, significant valvular disease, congenital heart disease, serious arrhythmia, stroke, or symptomatic peripheral artery disease (self-report, screening test)
  * Specific criteria used to determine whether a volunteer can undergo the screening CPET follow the American Heart Association (AHA) Criteria [54]
  * Inability to complete the CPET
  * Reassessment of the CPET may be allowed under some circumstances (e.g., test was not a maximal effort)
* Abnormal blood lipid profile (screening test)

  * Fasting triglycerides >500 mg/dL
  * Low-density lipoprotein cholesterol (LDL-C) >190mg/dL
* Cancer (self-report)

  * History of cancer treatment (other than non-melanoma skin cancer) and not "cancer-free" for at least 2 years
  * Anti-hormonal therapy (e.g., for breast or prostate cancer) within the last 6 months
* Chronic active or latent infection (self-report)

  * Active or latent infections requiring chronic antibiotic or anti-viral treatment
  * Chronic active infection whether on chronic antimicrobials or not
  * Human Immunodeficiency Virus
  * Active hepatitis B or C undergoing antiviral therapy
  * Individuals successfully treated for hepatitis C and virologically negative for at least 6 months are not excluded
* Liver enzyme tests (Alanine transaminase, Aspartate transaminase) (screening test)

  * >2 times the laboratory upper limit of normal
  * Reassessment during screening may be allowed under some conditions (e.g., recent use of acetaminophen)
  * Individuals may be referred to their PCP for evaluation; any medication change must be stable for ≥3 months prior to retesting
* Chronic renal insufficiency (screening test)

  * Estimated glomerular filtration rate <60 mL/min/1.73 m2 from serum creatinine (mg/dL) by the Chronic Kidney Disease Epidemiology Collaboration equation
  * Reassessment may be allowed under some conditions (e.g., questionable hydration status or other acute renal insult)
* Hematocrit (screening test)

  * Hematocrit >3 points outside of the local normal laboratory ranges for women and men
  * Reassessment may be allowed under certain conditions
  * Individuals may be referred to their PCP for evaluation; any medication change must be stable for ≥3 months prior to retesting
  * Individuals with known thalassemia trait may be included (despite having >3 points outside of the local normal laboratory ranges), upon approval from their PCP or a hematologist
* Blood donation (self-report)

  * Whole blood donation in the last 3 months or plans for blood donation during the entire protocol period
  * Platelet or plasma donation in the last week or plans for platelet or plasma donation during the entire protocol period
* Autoimmune disorders (self-report)

  * Individuals receiving any active treatment (including monoclonal antibodies) within the last 6 months
* Alcohol consumption (self-report)

  * More than 7 drinks per week for women
  * More than 14 drinks per week for men
  * History of binge drinking (≥5 drinks for males or ≥4 drinks for females in a 2-hour period more than once per month)
* Tobacco (self-report)

  * Current smokers: any tobacco or e-cigarette/e-nicotine products
  * Former smokers:
  * Stopped smoking <10 years at time of screening for those with a ≥20 pack-year smoking history
  * Stopped smoking <5 years at time of screening for those with a <20 pack-year smoking history
* Marijuana (self-report)

  * Self-reported use ≥3 days/week in any form
* Shift workers (self-report)

  * Night shift work in the last 6 months
  * Planning night shift work during the study period
* Cognitive status (screening)

  * Unable to give consent to participate in and safely complete the protocol, as based on the judgement of the local investigator
* Psychiatric illness (self-report and screening test)

  * Hospitalization for any psychiatric condition within one year (self-report)
  * Center for Epidemiological Studies-Depression Scale (CESD) score ≥16 [55] (screening test)
* Weight change (self-report)

  * Weight change (intentional or not) over the last 6 months of >5% of body weight
  * Plan to lose or gain weight during the study
* Lidocaine or other local anesthetic (self-report)

  * Known allergy to lidocaine or other local anesthetic
* COVID-19 infection

  * Hospitalization for COVID-19 infection in the past 12 months
  * Individuals who tested positive for COVID-19 but were not hospitalized must be symptom-free at least 14 days
* Other (clinician judgement)

  * Genetic metabolic disorders that could effect metabolomic results (e.g.,phenylketonuria)
  * Any other cardiovascular, pulmonary, orthopedic, neurologic, psychiatric. metabolic, or other conditions that, in the opinion of the local clinician, would preclude participation and successful completion of the protocol
  * Any other illnesses that, in the opinion of the local clinician, would negatively impact or mitigate participation in and completion of the protocol

EXCLUSIONS FOR MEDICATION USE

* Continuous use for 7 days or more of a new drug (prescription or over-the-counter; additional guidance in the MOP) in the last 3 months; eye and ear drops are allowed regardless of when they were started
* Dose change for any chronic-use drug in the last 3 months; changes in eye and ear drops are allowed
* Cardiovascular

  * Beta blockers and centrally acting anti-hypertensive drugs
  * Anticoagulants
  * Antiarrhythmic drugs
  * Antiplatelet drugs (other than aspirin ≤100 mg/day)
* Psychiatric drugs

  * Chronic use of medium or long-acting sedatives and hypnotics including all benzodiazepines; (short-acting non-benzodiazepine sedative-hypnotics are allowed)
  * Mood stabilizers
  * Antiepileptic drugs
  * Stimulants, Attention-Deficit/Hyperactivity Disorder (ADHD) drugs
  * Anti-psychotic drugs
* Pulmonary, inflammation

  * Chronic oral steroids; inhaled steroids are allowed
  * Burst/taper oral steroids more than once in the last 12 months; inhaled steroids are allowed
  * B2-agonists
  * allowed if on stable dose at least 3 months
* Genitourinary

  * 5-alpha reductase inhibitors
  * Daily phosphodiesterase type 5 inhibitor use
* Hormonal

  * Androgenic anabolic steroids
  * Anti-estrogens, anti-androgens
  * Estrogens and/or progestins used for reasons other than birth control or menopause
  * Growth hormone, insulin like growth factor-I, growth hormone releasing hormone
  * Any drugs used to treat diabetes mellitus or to lower blood glucose
  * Metformin for any indication
  * Any drugs used specifically to induce weight loss
  * Any drugs used specifically to induce muscle growth/hypertrophy or augment exercise-induced muscle hypertrophy
* Pain/inflammation

  * Narcotics and narcotic receptor agonists
  * Regular use of non-steroidal anti-inflammatory drugs (NSAIDs) or acetaminophen
  * Muscle relaxants ≥3 days per week
  * Oral/sublingual cannabidiol or similar in any formulation
* Other

  * Chronic systemic antimicrobials (antibiotic, antiviral, antifungal, antiparasite, etc) for any reason
  * High-potency topical steroids if ≥10% of surface area using rule of 9s
  * Continuous/chronic use of antibiotics or other anti-infectives for treatment or prevention
  * Monoclonal antibodies
  * Anti-rejection medications/immune suppressants
* Any other medications that, in the opinion of local clinicians, would negatively impact or mitigate full participation and completion

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1837 (Actual)
Dates: Start 2019-08-28 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Cardiopulmonary Exercise Test (CPET) VO2 Peak | Baseline; Week 12
  Changes in CPET VO2 Peak calculated as L/min
Isometric Knee Peak Torque by Group | Baseline; Week 12
  Changes in peak torque measured in Newton Meters

SECONDARY OUTCOMES:
HDL-C | Baseline; Week 12
  Changes in HDL-C (mg/dL)
LDL-C | Baseline; Week 12
  Changes in LDL-C (mg/dL)
Triglycerides | Baseline; Week 12
  Changes in Triglycerides (mg/dL)
HbA1C | Baseline; Week 12
  Changes in HDL-C (mg/dL)

CONTACTS AND LOCATIONS:
Overall Officials: Mike E Miller, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (11):
- United States (11):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of Colorado Denver, Denver, Colorado
  - Florida Hospital / Advent Health, Orlando, Florida
  - Ball State University, Muncie, Indiana
  - Pennington Biomedical Research Center, Baton Rouge, Louisiana
  - Duke University Medical Center, Durham, North Carolina
  - East Carolina University, Greenville, North Carolina
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Texas Medical Branch - Galveston, Galveston, Texas
  - University of Texas Health Science Center, San Antonio, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared publicly through the MoTrPAC data hub based on the consent and assent choices of the parent/participant. PHI will not be released.
Supporting Information: Study Protocol
Time Frame: The timeframe for data sharing is unknown at this time. Estimated time for release is end of 2026.
Access Criteria: All data and supporting information will be made available through the MoTrPAC Data Hub (https://motrpac-data.org/). Data Access can be requested and public repositories will be outlined on the data hub website.
URL: https://motrpac-data.org/

REFERENCES:
- [Background] MoTrPAC Study Group; Jakicic JM, Kohrt WM, Houmard JA, Miller ME, Radom-Aizik S, Rasmussen BB, Ravussin E, Serra M, Stowe CL, Trappe S, Abouassi H, Adkins JN, Alekel DL, Ashley E, Bamman MM, Bergman BC, Bessesen DH, Broskey NT, Buford TW, Burant CF, Chen H, Christle JW, Clish CB, Coen PM, Collier D, Collins KA, Cooper DM, Cortes T, Cutter GR, Dubis G, Fernandez FM, Firnhaber J, Forman DE, Gaul DA, Gay N, Gerszten RE, Goodpaster BH, Gritsenko MA, Haddad F, Huffman KM, Ilkayeva O, Jankowski CM, Jin C, Johannsen NM, Johnson J, Kelly L, Kershaw E, Kraus WE, Laughlin M, Lester B, Lindholm ME, Lowe A, Lu CJ, McGowan J, Melanson EL, Montgomery S, Moore SG, Moreau KL, Muehlbauer M, Musi N, Nair VD, Newgard CB, Newman AB, Nicklas B, Nindl BC, Ormond K, Piehowski PD, Qian WJ, Rankinen T, Rejeski WJ, Robbins J, Rogers RJ, Rooney JL, Rushing S, Sanford JA, Schauer IE, Schwartz RS, Sealfon SC, Slentz C, Sloan R, Smith KS, Snyder M, Spahn J, Sparks LM, Stefanovic-Racic M, Tanner CJ, Thalacker-Mercer A, Tracy R, Trappe TA, Volpi E, Walsh MJ, Wheeler MT, Willis L. Molecular Transducers of Physical Activity Consortium (MoTrPAC): human studies design and protocol. J Appl Physiol (1985). 2024 Sep 1;137(3):473-493. doi: 10.1152/japplphysiol.00102.2024. Epub 2024 Apr 18. PMID 38634503

DOCUMENTS (1):
  • Informed Consent Form (2025-02-18): https://cdn.clinicaltrials.gov/large-docs/27/NCT03960827/ICF_000.pdf